CLINICAL TRIAL: NCT02560519
Title: Albumin vs Ringer Solution for Cardiac Surgery
Brief Title: Albumin in Cardiac Surgery
Acronym: ALBICS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Maxim Mazanikov, Dr, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPA1
Record Dates: First submitted 2015-09-24; First posted 2015-09-25 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: C.Surgical Procedure; Cardiac
Keywords: human serum albumin solution; Cardiopulmonary Bypass
MeSH Terms: interventions — Albumins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ringers acetate solution (Active Comparator): Ringer-Acetat Baxter Viaflo® (Baxter Finland, Finland): Ringer-Acetat is iso-oncotic solution.Pharmacodynamic and pharmacokinetic properties: The osmotic effect is approximately the same as that of blood plasma. Electrolytes are given to receive or to keep normal osmotic conditions in the extracellular as well as the intracellular compartment. Acetate is oxidized into bicarbonate, mainly in the muscles and peripheral tissues and gives a weak alkalizing effect. Qualitative and quantitative list of composition: 1000 ml of Ringer-Acetat Baxter Viaflo contains 5.86 g sodium chloride, 0.30 g potassium chloride dihydrate, 0.29 g, 0.20 g magnesium chloride hexahydrate, 4.08 g sodium acetate trihydrate. List of excipients: Water for injections, Hydrochloric acid.
  Interventions: Drug: Ringers acetate solution
- Albumin solution (Experimental): Albuman® 200g/L (Sanquin, the Netherlands) is a solution containing 200 g/l (20%) of total protein of which at least 95% is human albumin.The solution contains 100 mmol/l of sodium (2.3 g/L). Pharmacodynamic properties: Albumin stabilises circulating blood volume and is a carrier of hormones, enzymes, medicinal products and toxins. Pharmacokinetic properties. Under normal conditions, the average half-life of albumin is about 19 days. Albuman® 40g/L is a solution containing 40 g/l (4%) of total protein of which at least 95% is human albumin. The solution contains 140 mmol/l of sodium (3.2 g/L).
  Interventions: Drug: Albumin solution

INTERVENTIONS:
Drug: Albumin solution — Albumin solution will used for priming of the CPB(cardio-pulmonary bypass) tubing. : A mixture of 20% (200 mg/mL) albumin (Albuman® 200 g/L, Sanquin, the Netherlands) with Ringer's acetate solution in the final albumin concentration of 4%.
  During surgery and the first 24 hours of ICU treatment, albumin 4% solution will be used up to 3200 mL for volume replacement therapy. Ringer's acetate solution is used thereafter, i.e. if more than 3200 mL are needed for volume replacement therapy.The volume replacement therapy is not determined but will be based on the clinical decision.
  Other Names: Albumin
  Arms: Albumin solution
Drug: Ringers acetate solution — The Ringers acetate solution will be used for priming of the CPB tubing. The CPB priming volume comprises only of Ringer´s solution.
  During surgery and the first 24 hours of ICU treatment,Ringer´s acetate solution will be used up to 3200 mL for volume replacement therapy. Ringer's acetate solution is used thereafter, i.e. if more than 3200 mL are needed for volume replacement therapy during the second study phase. The volume replacement therapy is not determined but will be based on the clinical decision.
  Arms: Ringers acetate solution

SUMMARY:
Colloid solutions are widely used for volume replacement therapy because of their high oncotic pressure, which could reduce interstitial fluid shifting. Human albumin is the only colloid solution of biologic origin with a molecular weight of 60 kDa. As the most abundant plasma protein, it has physiological importance in the well-being of the endothelial glycocalyx. Older studies in septic patients, however, did not show any benefit of albumin over saline solution. Crystalloid solutions, such as Ringer's acetate, do not impair neither renal function nor coagulation, but their volume expanding effect is questionable.

For several reasons (use of heart-lung machine, systemic inflammation, coagulation disturbances), patients undergoing cardiac surgery need especially large amounts of fluids. However, there are no large trials comparing albumin solutions to crystalloid solutions cardiac surgery.

This double-blinded trial will randomize according to a power analysis 1250 cardiac surgery patients (=625+625) at Meilahti hospital to use either 4% Albumin or Ringer's acetate solutions for both priming of the heart-lung machine and perioperative volume replacement therapy. The primary efficacy and safety endpoint of this study is the incidence of major adverse events (MAE), defined as a composite endpoint of all-cause mortality, acute myocardial infarction, acute heart failure or low output syndrome, resternotomy, stroke, certain arrhythmias, major bleeding, infections compromising post-procedural rehabilitation, acute kidney injury within 90 days postoperatively. The secondary outcomes are total number of MAEs, major adverse cardiac events (MACE), perioperative fluid balance, blood product transfusions, blood loss, acute kidney injury, days alive without mechanical ventilation/outside ICU/at home in 90 days as well as 90-day mortality. Blood samples for biochemical analyses will be collected at four perioperative time points.

This trial will provide data about efficacy and safety of 4% albumin in cardiac surgery patients. The biochemical mechanisms of albumin will be assessed.

DETAILED DESCRIPTION:
The use of cardiopulmonary bypass (CPB) between two study solutions: albumin solution with the final concentration of 4% and Ringer's acetate solution. The trial consists of two phases as follows. For each patient, one and the same study solution will used in both phases of the trial according to randomization.

In the first phase of the trial, the study solution will be used for priming of the CPB tubing. The CPB priming volume comprises only of the study solution. See the Blinding section below for more details.

* Albumin group (trial group): A mixture of 20% (200 mg/mL) albumin solution (Albuman® 200 g/L, Sanquin, the Netherlands) with Ringer's acetate solution (see below) in the final albumin concentration of 4%.
* Ringer group (conventional group): Ringer's acetate solution (Ringer-acetate®, Baxter; pH 6.0, contents Na+ 131 mmol/L, Cl- 112 mmol/L, acetate 30 mmol/L) alone.

In the second phase of the trial, during surgery and the first 24 hours of ICU treatment, study solution will be used up to 3200 mL for volume replacement therapy. Ringer's acetate solution is used thereafter, i.e. if more than 3200 mL are needed for volume replacement therapy during the second study phase. The volume replacement therapy is not protocolled but will be based on the clinical decision.

Albumin group (trial group):4% (40 mg/mL) albumin(Albuman®, Sanquin, the Netherlands)

•Ringer group (conventional group): Ringer's acetate solution (Ringer-acetate®, Baxter; pH 6.0, contents Na+ 131 mmol/L, Cl- 112 mmol/L, acetate 30 mmol/L) The trial will end after the first 24 hours of ICU treatment or when the patient leaves the ICU if the latter occurs within the first postoperative 24 hours. After the study period, fluids are administered according to the local clinical practice.

The use of blood products, excluding albumin, is not protocolled, but will be based on the clinical decision.

For physiological basic need of fluid, Ringer's acetate solution will be given throughout the study period, i.e. during surgery and postoperatively, as a background infusion of 0.5 ml/kg/h, rounded to the nearest multible of 10 ml.

ELIGIBILITY:
Inclusion Criteria:

* following primary or repeat open heart surgery procedures, either independently or in combinations:CABG,aortic valve replacement/repair, mitral valve replacement/repair,tricuspid valve replacement/repair,the MAZE procedure or its modifications,surgery on the aortic root or ascending aorta not requiring hypothermic circulatory arrest;
* scheduled for elective surgery or operated during the index admission

Exclusion Criteria:

* immediate emergency surgery (i.e. no time for recruitment)
* end-stage kidney disease (estimated GFR<20 mL/min - based on serum/ plasma creatinine)
* hemophilia A, hemophilia B
* patient denial of the use of blood products and derivatives of blood products
* ticagrelor, prasugrel, clopidogrel,apixaban or rivaroxaban treatment within 2 days preoperatively or that of dabigatran within 3 days
* correction of a congenital heart defect
* preoperative infection compromising post-procedural rehabilitation
* preoperative heart failure / low output syndrome (preoperative inotropic support, intra-aortic balloon pump, preoperative EF(ejection fraction) < 20 %)
* preoperative dependency of mechanical ventilation, preoperative ECMO(extra-corporeal membrane oxygenation),left ventrical mechanical assistance.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1386 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
Major adverse events | 90 days
  The number of patients with at least one major adverse event during 90 days postoperatively:all-cause death;acute myocardial injury (increase in CK-MB at least 10 times as high as the upper normal limit);new onset of acute heart failure/low output syndrome requiring intravenous inotropic agents,intra-aortic balloon pump support and/or ECMO,resternotomy/subxiphoidal pericardial drainage;stroke;major arrhythmia (ventricular fibrillation off-CPB,ventricular tachycardia off-CPB,new onset atrial fibrillation of permanent nature requiring anticoagulation, permanent pacing dependency of new onset);major bleeding (chest tube blood loss at 18 hours over 20 mL/kg) or requiring 5 or more units of red blood cell transfusion or an equivalent volume of washed red blood cells within intervention time;infection compromising post-procedural rehabilitation;acute kidney injury(postoperative increase of creatinine at least 2 times compared to the preoperative level),renal replacement therapy

CONTACTS AND LOCATIONS:
Overall Officials: Eero Pesonen, MD.,PhD, Study Chair — Helsinki University Central Hospital; Hanna Vlasov, MD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Meilahti Hospital, Helsinki, Uusimaa, Finland

REFERENCES:
- [Derived] Pesonen E, Vlasov H, Suojaranta R, Hiippala S, Schramko A, Wilkman E, Eranen T, Arvonen K, Mazanikov M, Salminen US, Meinberg M, Vahasilta T, Petaja L, Raivio P, Juvonen T, Pettila V. Effect of 4% Albumin Solution vs Ringer Acetate on Major Adverse Events in Patients Undergoing Cardiac Surgery With Cardiopulmonary Bypass: A Randomized Clinical Trial. JAMA. 2022 Jul 19;328(3):251-258. doi: 10.1001/jama.2022.10461. PMID 35852528
- [Derived] Vlasov H, Juvonen T, Hiippala S, Suojaranta R, Peltonen M, Schramko A, Arvonen K, Salminen US, Kleine Budde I, Eranen T, Mazanikov M, Meinberg M, Vahasilta T, Wilkman E, Pettila V, Pesonen E. Effect and safety of 4% albumin in the treatment of cardiac surgery patients: study protocol for the randomized, double-blind, clinical ALBICS (ALBumin In Cardiac Surgery) trial. Trials. 2020 Feb 28;21(1):235. doi: 10.1186/s13063-020-4160-3. PMID 32111230